CLINICAL TRIAL: NCT01603160
Title: Improving Emergency Department Management of Adults With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Wake Forest University Health Sciences (Other); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00032162; 1R18HS019646-01A1 (AHRQ)
Record Dates: First submitted 2012-04-16; First posted 2012-05-22 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Emergency Department; Quality Improvement
MeSH Terms: conditions — Anemia, Sickle Cell; Emergencies | interventions — Quality Improvement

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Emergency Department Staff: Interventions put in place in the Emergency Department will effect most staff who work in the ED, but different sub-groups will be approached for participation in specific aspects of the study:
  * All ED attending and resident physicians and ED nurses will be invited to complete the SCD Attitudes survey.
  * Select ED Staff will be invited to be members of the QI team and will be invited to participate in the FMECA.
  * Members of the QI team will be invited to participate in a focus group.
  Interventions: Behavioral: Quality Improvement

INTERVENTIONS:
Behavioral: Quality Improvement — There are no interventions for the individual patient. The changes in processes developed by the quality improvement team will be made for all adults with sickle cell disease, not just adults who consent to interviews.
  A proactive risk assessment methodology, Failure Modes, Effects, and Criticality Analysis (FMECA), will be used in two EDs to identify the vulnerabilities, risks, and weak points (failures) in the systems and processes involved in four key decisions of the ED-SCANS. Based on the aggregated results of the FMECA's, generalizable quality improvement interventions (QII's) will be developed and implemented with the purpose of changing the way emergency care for adults with SCD is delivered and organized.

SUMMARY:
The objective of this study is to design, implement and test quality improvement measures to improve the care of adults with sickle cell disease in the emergency department.

DETAILED DESCRIPTION:
There is a critical need to consistently provide best practice care for adult patients with sickle cell disease (SCD) who present to emergency departments (EDs). Patients with SCD suffer a shortened lifespan, and often die of many disease associated complications in their 4th and 5th decade of life. These complications include, but are not limited to: stroke, sepsis, pulmonary embolus, acute chest syndrome, and multi-system organ failure. Patients typically present to the ED with severe acute pain that requires rapid analgesic administration, often with high doses of opioids. The perception among many clinicians is that these patients, usually African American, are "drug seeking". This results in delays to administration of analgesics and inferior pain management. Finally, a small proportion of adults with SCD have a large number of visits. A recent study revealed that approximately 25% of adult patients with SCD had more than six ED visits per year with about 10% having more than 23 visits. Several patients had up to 175 visits over a 2-year period. There is also evidence that SCD patients with more than two hospitalizations/year are at an increased risk of death. ED clinicians are often frustrated when they see the same patient for multiple ED visits. This also leads to inadequate analgesic management. These issues highlight the suboptimal effectiveness of the process and systems of ED care for adults with SCD. ED practices for SCD care would significantly benefit from re-design and implementation of innovative best practice management strategies to optimize ED evaluation and management of VOC-related pain and facilitate appropriate referral to a primary care provider.

The ED-SCANS is a validated and reliable decision support tool developed by the principal investigator to help guide ED clinicians in delivering best practice care to adults with SCD. However, optimal integration of the tool within ED systems and process of care and the effect of the tool on both ED system and patient outcomes have not been evaluated. This study is the next logical step in the implementation of the ED-SCANS. The proposed study will use four key decisions of the ED-SCANS (triage, analgesic management, identification of high risk patients, and patient referral for care) as a framework to improve the processes and systems in ED management of adults with SCD. A proactive risk assessment methodology -- Failure Modes, Effects, and Criticality Analysis (FMECA) -- will be used in two EDs to identify the vulnerabilities, risks, and weak points (failures) in the systems and processes involved in four key decisions of the ED-SCANS. Based on the aggregated results of the FMECA's, generalizable quality improvement interventions (QII's) will be developed and implemented with the purpose of changing the way emergency care for adults with SCD is delivered and organized. These re-designed systems and processes (interventions) will be developed to be generalizable to most EDs, with minor modifications. A formal program evaluation will be conducted to determine the barriers and facilitators to implementation of the interventions. Preliminary, hypothesis generating data will be collected for selected outcomes related to each of the four decisions associated with the ED-SCANS. A toolbox of educational materials and electronic medical record prompts for EDs will be developed to facilitate implementation of the ED-SCANS at EDs across the country. This study will therefore focus on (1) developing an optimal implementation strategy using formal risk assessment (FMECA) and quality improvement (PDSA) methods focused on four key decisions of the ED-SCANS: Decision 1: triage, Decision 2: analgesic management, Decision 3: identification of high risk patients, and Decision 7: patient referral for care to improve the processes and systems involved in the care of adults with SCD and (2) conducting a formal program evaluation consisting of a process evaluation (to understand whether the optimal implementation strategy performs as intended (e.g. actual versus planned) through assessment of the barriers and facilitators to the implementation) and an outcomes evaluation of relevant clinical performance indicators, and patient and clinician outcomes. The outcome evaluation is designed to be hypothesis generating, not hypothesis testing. Finally, a toolbox of educational materials and other implementation tools such as decision support tools (e.g., documentation templates) will be developed during the project.

ELIGIBILITY:
Inclusion Criteria for Patient Subjects:

* 18 years and older
* Ability to read and understand English
* Diagnosis of Sickle Cell Disease

Exclusion Criteria for Patient Subjects:

* Diagnosis of Sickle Cell Trait, vs. Disease

Inclusion Criteria for Clinician Subjects:

* Attending or resident physician, or nurse in the Emergency Department

Exclusion Criteria for Clinician Subjects:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient subjects will be recruited from the Duke University and Wake Forest Emergency Departments. All ED attending and resident physicians and ED nurses will be invited to complete the SCD Attitudes survey. Ten clinicians at Duke and 10 clinicians at Wake Forest will be recruited to participate in the FMECA's.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of SCD patients meeting high user criteria | 3, 6, 9, 12, 15, 18, 21, 24, and 27 months
  High user criteria include: No Primary Care Physician, >3 painful episodes per year, >3 ED visits or hospitalizations per year, difficulty getting appointments with PCP. Specific outcome measures include: decrease in the number of ED visits and hospitalizations, as well as improvement in the proportion of physician, social service, and psychiatric service referrals made for high risk/high utilizer patients when indicated. Data will be collected via quarterly medical record reviews (every quarter) and patient interviews (quarters 3-10).
Change in clinical performance indicators and patient and clinician outcome measures | 3, 6, 9, 12, 15, 18, 21, 24, and 27 months
  This outcome is exploratory and designed to be hypothesis generating. A combination of clinical performance indicators and patient and clinician outcomes will be analyzed, including Triage Score (correct/incorrect), Time to initial analgesic from arrival (minutes from arrival to administration of 1st dose), and patient satisfaction with ED analgesic management.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, MSN, MPH, PhD, RN, Principal Investigator — Duke University
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States